CLINICAL TRIAL: NCT03211910
Title: Sacral Savers: Study of Prevention and Enhanced Healing of Sacral and Trochenteric Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issue of the sponsor
Sponsor: Richmond University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-04-11
Record Dates: First submitted 2017-06-01; First posted 2017-07-07 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Healing Ulcer
Keywords: Sacral and trochenteric pressure ulcers

STUDY DESIGN:
Intervention Model Description: Sacral Savers is a combination of a strong bubble wrap sheet with a fold at the head end and a nylon sham with a pocket into which the bubble wrap sheet is inserted. This combination is then placed under the fitted sheet on the patient's • Intervention:: medical device: Bubble wrap mattress has been successful in enhancing wound healing. Wound healing is greater than 20% healing within two weeks documented by measurement of the wound bed or wound healing to less than the dermal layer documented by photography and agreement of healing between research associate and physician . The bubble wrap mattress will be place underneath the participant. Follow-up will occur weekly for 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Care of Treatment (Placebo Comparator): Participants will be treated with standard of care treatment.
  Interventions: Other: Standard Care of Treatment
- SacralSaver (Active Comparator): SacralSaver
  Interventions: Device: SacralSaver

INTERVENTIONS:
Device: SacralSaver — Sacral Savers is a combination of a strong bubble wrap sheet with a fold at the head end and a nylon sham with a pocket into which the bubble wrap sheet is inserted. This combination is then placed under the fitted sheet on the patient's mid back and the pressure exerted by the lower back of the patient is markedly reduced or nearly eliminated (tested and proven using computer models), thereby preventing the onset of pressure ulcers in the sacro-coccygeal area.
  Arms: SacralSaver
Other: Standard Care of Treatment — Standard Care of Treatment
  Arms: Standard Care of Treatment

SUMMARY:
The purpose of the study is to investigate the ability of the product "Sacral Saver," to prevent and /or help healing bed sores.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate the ability of the product "Sacral Savers." to prevent and/or help healing of bed sores, in patients in health care facilities.

The Sacral saver device consists of a sheet of strong bubble-wrap-like material, folded at one end and covered by a nylon sham with a pocket in which the bubble wrap is placed. The assembled device is placed under the bed sheet in such a way that the small of the back rests on the fold. This will lift the back and reduce the pressure of the buttocks on the bed. When lying on the side, it will reduce the pressure on the hip.

Participants are being asked to participate in this study because you are at risk for, or already have a bedsore on the buttocks or the hip.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is immobilized for prolonged periods, either in acute care, or chronic care situations.
* All patients with: paralysis, quadriplegia, paraplegia, trauma patients, requiring prolonged immobilization, patients on ventilators.
* All patients with pre-existing pressure ulcers in the lower back and or hip regions.

Exclusion Criteria:

* There are no age, gender or co-morbidity exclusions

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Bubble wrap mattress for Pressure Ulcer prevention, measured by a ruler (cm) | 6 weeks
  This pilot study of 30 participants (15 control, 15 experimental) will test the safety and efficacy of using a bubble wrap mattress for pressure ulcer. Participants in one group would receive standard of care treatment and the other group would receive the intervention of the bubble wrap mattress. Participants would be followed for 6 weeks to assess wound healing and tolerance of the treatment. of ulcers. The outcome measure will measure 30 participants, 15 treated with the SacralSavers device and 15 participants with standard of care treatment up to the resolution of the participant's ulcer.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis A Bloomfield, MD, Principal Investigator — Richmond University Medical Center
Locations (1):
- Richmond University Medical Center, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bluestein D, Javaheri A. Pressure ulcers: prevention, evaluation, and management. Am Fam Physician. 2008 Nov 15;78(10):1186-94. PMID 19035067
- [Background] Macon L, Sloan M, What you should know about decubitus ulcers. November 2015
- [Background] Reddy M, Gill SS, Rochon PA. Preventing pressure ulcers: a systematic review. JAMA. 2006 Aug 23;296(8):974-84. doi: 10.1001/jama.296.8.974. PMID 16926357
- [Background] Medical Advisory Secretariat. Management of chronic pressure ulcers: an evidence-based analysis. Ont Health Technol Assess Ser. 2009;9(3):1-203. Epub 2009 Jul 1. PMID 23074533
- [Background] Kirman CN.Pressure ulcer and wound care.Medscape.June 2016